CLINICAL TRIAL: NCT03193177
Title: A Retrospective and Prospective Cohort Study of the 21-day Fasting-like Diet in Patients With Metabolic and Autoimmune Diseases
Status: Completed | Type: Observational
Sponsor: Tsinghua University (Other)
Collaborators: Nanshan Branch of Qilu Hospital (Unknown)
Responsible Party: Principal Investigator, Minghui Zhang, Associate Professor, Tsinghua University
Other Study IDs: THUMED-BG-170612
Record Dates: First submitted 2017-06-12; First posted 2017-06-20 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Fasting; Chronic Disease; Autoimmune Diseases; Metabolic Disease; High Blood Pressure; Fatty Liver; Kidney Stone; Gall Stone; Hysteromyoma
Keywords: fasting-like diet; chronic diseases; autoimmune diseases; metabolic disorder
MeSH Terms: conditions — Fasting; Chronic Disease; Autoimmune Diseases; Metabolic Diseases; Hypertension; Fatty Liver; Kidney Calculi; Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the 21-day fasting-like diet: Participants will be supplied with fasting-like diet containing only 5% of normal calorie intake. Physical examinations will be performed on day 0, 4,7,14,21 and 51 after the clinical trial.
  Interventions: Other: the 21-day fasting-like diet

INTERVENTIONS:
Other: the 21-day fasting-like diet — a fasting-like diet with 400 KJ energy intake per day for 21 days
  Other Names: Bigu

SUMMARY:
Effectiveness of fasting or fasting-mimicking diet has been proved an effective approach to treat metabolic and autoimmune diseases in mice. However, clinical trials performing prolonged fasting with more than 7 days have not been reported. Investigators conduct an open label, phase I/II clinical trial to evaluate the safety and effectiveness of the 21-day fasting-like diet in the treatment of metabolic and autoimmune diseases.

DETAILED DESCRIPTION:
Although fasting has been proved an effective approach to treat metabolic and autoimmune diseases in mice, prolonged fasting is difficult to implement in human-beings for the safety and feasibility reasons.

In this clinical trial, we will recruit metabolic and autoimmune diseases and then follow a traditional Chinese 21-day fasting-like diet process with extremely low calorie intake (about 5% of normal diet) and prolonged fasting-like period. Blood, urine, stool samples will be collected on day 0 (baseline), day 4, day 7, day 14, day 21 and day 51 after it started up. Therefore we can examine the changes of disease-associated physical indexes and metabolic biomarkers pre and post the 21-day fasting-like diet.

The purpose of the study is to ascertain the impact of the fasting-like diet during the 21 days. The investigators hypothesize that the 21-day fasting-like diet can reduce the biomarkers associated with aging and age-related diseases and benefit for the treatment of metabolic and autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥18 and ≤75 years;
* Subjects has a confirmed diagnosis of metabolic and autoimmune diseases, including high blood pressure, kidney stone, gall stone, hysteromyoma, fatty liver, psoriasis, and so on.

Exclusion Criteria:

* Subjects has a confirmed diagnosis of cancer;
* Females who are pregnant or nursing;
* Subject requires a prescheduled regularly administration of drugs;
* Subject has severe renal insufficiency;
* Subject has cardiac arhythmia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Of these 144 participants, 55 were male and 89 were female. For detailed information, please follow our recent publications.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 30 days after the fasting-like diet
  Phase I: To obtain preliminary estimates of the safety of the fasting-like diet.
Evaluation of the therapeutic effects on metabolic disorder-associated diseases by the examination of metabolic biomarkers. | 30 days after the fasting-like diet
  Phase II: To compare the state of diseases pre and post fasting-like diet by the examination of comprehensive metabolic panel.

SECONDARY OUTCOMES:
Functional changes in the peripheral blood lymphocytes pre and post fasting-like diet as accesse by flow cytometry and RNA-seq. | Baseline, 4 days, 7 days, 14 days, 21 days, 51 days after the beginning of the fasting-like diet
  Peripheral blood samples were collected at indicated time points and analyzed by flow cytometry for the composition of lymphocyte subsets and by RNA-seq for their functions.
Compositional changes in intestinal microflora pre and post fasting-like diet as accesse by RNA-seq. | Baseline, 4 days, 7 days, 14 days, 21 days, 51 days after the beginning of the fasting-like diet
  Stool samples were collected in time if possible and analyzed by RNA-seq for the composition of the intestinal microflora.

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Ming, MD, Study Director — Nanshan Branch of Qilu Hospital
Locations (1):
- Nanshan Branch of Qilu Hospital, Longkou, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes